CLINICAL TRIAL: NCT01664819
Title: Antioxidants for Prevention of Cataracts Follow-up Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Aravind Eye Hospitals, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: P0047247
Record Dates: First submitted 2012-08-10; First posted 2012-08-14 (Estimated); Last update posted 2018-10-30 (Actual); Status verified 2018-10

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract | interventions — Antioxidants

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Antioxidant supplementation (Active Comparator): Randomized to receive antioxidant supplementation (vitamin C, 500 mg; beta carotene, 15 mg; and alpha-tocopherol, 400 IU) three times per week for five years.
  Interventions: Dietary Supplement: Antioxidant
- Placebo (Placebo Comparator): Randomized to receive placebo three times per week for five years
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Antioxidant
  Arms: Antioxidant supplementation
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
Aravind Eye Hospital and the University of California, San Francisco (UCSF) Proctor Foundation collaborated on the Antioxidants for the Prevention of Cataract Study from 1997-2002. (1) In the study, 798 participants aged 35-50 years were enrolled from 5 rural villages, and randomized to thrice weekly antioxidants (vitamin C, 500 mg; beta carotene, 15 mg; and alpha-tocopherol, 400 IU) or placebo. After 5 years of supplementation, there was no significant difference in cataract formation between the antioxidant group and placebo. In this follow-up study, we will return to study villages to determine whether rates of cataract surgery are different in the 2 groups.

1. Gritz DC, Srinivasan M, Smith SD, et al. The Antioxidants in Prevention of Cataracts Study: effects of antioxidant supplements on cataract progression in South India. The British journal of ophthalmology 2006;90:847-51.

ELIGIBILITY:
Inclusion Criteria:

* participation in previous cataract study

Exclusion Criteria:

* refusal to participate

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 576 (Actual)
Dates: Start 2012-08; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Cataract surgery | 15 years post-intervention
  Effect of intervention on cataract surgery 15 years post-intervention in a logistic regression model

SECONDARY OUTCOMES:
Risk factors for cataract surgery | 15 years post-intervention
  Association of risk factors assessed via questionnaire 15 years ago with cataract surgery in a multiple logistic regression model
All-cause mortality | 15 years post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy D Keenan, MD, MPH, Principal Investigator — University of California, San Francisco; Muthiah Srinivasan, MD, Principal Investigator — Aravind Eye Hospitals
Locations (1):
- Aravind Eye Hospitals, Madurai, Tamil Nadu, India

REFERENCES:
- [Background] Gritz DC, Srinivasan M, Smith SD, Kim U, Lietman TM, Wilkins JH, Priyadharshini B, John RK, Aravind S, Prajna NV, Duraisami Thulasiraj R, Whitcher JP. The Antioxidants in Prevention of Cataracts Study: effects of antioxidant supplements on cataract progression in South India. Br J Ophthalmol. 2006 Jul;90(7):847-51. doi: 10.1136/bjo.2005.088104. Epub 2006 Mar 23. PMID 16556618
- [Derived] Nesemann JM, Srinivasan M, Ravindran RD, Edwards T, O'Brien KS, Kim UR, Wilkins JH, Whitcher JP, Lietman TM, Gritz DC, Keenan JD. Relationship Between Cooking Fuel and Lens Opacities in South India: A 15-Year Prospective Cohort Study. Am J Ophthalmol. 2022 Nov;243:66-76. doi: 10.1016/j.ajo.2022.06.021. Epub 2022 Jul 9. PMID 35817091